CLINICAL TRIAL: NCT06986590
Title: Addressing Hypertension Care in Africa (ADHINCRA) Program
Brief Title: Addressing Hypertension Care in Africa Program
Acronym: ADHINCRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00504718; 1R01HL175642-01 (NIH)
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Hypertension; High Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Stepped wedge cluster randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): This cohort will be the first to participate in the ADHINCRA Program, which includes home blood pressure monitoring, an mHealth app, nurse-led lifestyle counselling and treatment with a simplified hypertension control protocol.
  Interventions: Behavioral: ADHINCRA Program
- Cohort 2 (Experimental): This cohort will begin the ADHINCRA Program 3 months after Cohort 1.
  Interventions: Behavioral: ADHINCRA Program
- Cohort 3 (Experimental): This cohort will begin the ADHINCRA Program 6 months after Cohort 1.
  Interventions: Behavioral: ADHINCRA Program
- Cohort 4 (Experimental): This cohort will begin the ADHINCRA Program 9 months after Cohort 1.
  Interventions: Behavioral: ADHINCRA Program

INTERVENTIONS:
Behavioral: ADHINCRA Program — The ADHINCRA Program is a nurse-led intervention that includes the use of home blood pressure monitoring, a mobile health app, lifestyle counselling, and a simplified hypertension treatment protocol to achieve blood pressure control among people diagnosed with hypertension.

SUMMARY:
The ADHINCRA Program is a bundle of multilevel evidence-based interventions that address multiple predictors of controlled hypertension, including patient-, provider-, and health system-level factors. The successful implementation of the ADHINCRA program will provide a rigorous and scalable model for improving hypertension control in Africa, which would ultimately reduce the risk of cardiovascular disease, stroke and kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 -70 years.
* Diagnosis of hypertension and elevated systolic blood pressure measure (≥140 mmHg) on the most recent clinic visit without a diabetes diagnosis.
* Hypertension treatment naive or on monotherapy.
* Receives primary care at one of the participating sites.
* Willing and able to provide informed consent in English, Twi, Dagbani, Ewe, Hausa, or Yoruba.
* Owns a smartphone (Android or iOS).

Exclusion Criteria:

* Age <18 years or >70 years.
* Severely elevated BP (≥180/110mmHg).
* Diagnosis of stroke, coronary artery disease, or kidney disease.
* Diagnosis of end-stage renal disease (ESRD) treated with dialysis.
* Serious medical condition which either limits life expectancy or requires active management (e.g., cancer).
* Cognitive impairment or other conditions preventing study participation
* Pregnant or currently nursing a child
* Unwilling to provide informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with systolic blood pressure <140 mmHg | Baseline and 12 months post-randomization
  Blood pressure control among participants defined as systolic blood pressure <140 mmHg

SECONDARY OUTCOMES:
Number of participants with diastolic blood pressure <90 mmHg | Baseline, 12 months, 24 months post-randomization
  Blood pressure control as assessed by diastolic blood pressure <90mmHg
Medication adherence as assessed by Hill-Bone Medication Adherence Scale | Baseline, 12 months, 24 months post-randomization
  Adherence to medications prescribed per the ADHINCRA Program treatment protocol. The total score ranges from 14 - 56. Higher score is better adherence.
Percentage of sites that adopt and maintain the intervention as assessed by the Pragmatic Robust Implementation and Sustainability Model | Baseline, 12 months, 24 months post-randomization
  Use the Pragmatic Robust Implementation and Sustainability Model (PRISM) to evaluate the reach, adoption, maintenance of the ADHINCRA Program
Difference in cost of intervention compared to usual care as assessed by the Pragmatic Robust Implementation and Sustainability Model | Baseline, 12 months, 24 months post-randomization
  Use the Pragmatic Robust Implementation and Sustainability Model (PRISM) to evaluate the cost-effectiveness of the ADHINCRA Program

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Commodore-Mensah, PhD, MHS, RN, Principal Investigator — Johns Hopkins University; Fred S Sarfo, MBBS, PhD, FWACP, Principal Investigator — Kwame Nkrumah University of Science and Technology; Dike B Ojji, MBBS, PhD, FWACP, Principal Investigator — University of Abuja
Locations (17):
- Johns Hopkins University, Baltimore, Maryland, United States
- Ghana (10):
  - Dominase SDA Hospital, Bekwai, Ashanti Region
  - Kumasi South Hospital, Kumasi, Ashanti Region
  - Manhyia Government Hospital, Kumasi, Ashanti Region
  - Tafo Government Hospital, Tafo, Ashanti Region
  - Berekum Holy Family Hospital, Berekum, Bono
  - St. John of God Catholic Hospital, Duayaw Nkwanta, Bono
  - Northern Regional Hospital, Tamale, Northern Region
  - Tamale Teaching Hospital, Tamale, Northern Region
  - Ho Municipal Hospital, Ho, Volta Region
  - South Tongu District Hospital, Sogakope, Volta Region
- Nigeria (6):
  - Akure South Hospital, Akure, Ondo State
  - Akoko North East, Ondo, Ondo State
  - Akoko North West, Ondo, Ondo State
  - Akoko South East, Ondo, Ondo State
  - Akoko South West, Ondo, Ondo State
  - Owo General Hospital, Owo, Ondo State

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Commodore-Mensah Y, Sarfo FS, Turkson-Ocran RA, Foti K, Mobula LM, Himmelfarb CD, Carson KA, Appiah LT, Degani M, Lang'at C, Nyamekye G, Molello NE, Ahima R, Cooper LA. Addressing Hypertension Care in Africa (ADHINCRA): Study protocol for a cluster-randomized controlled pilot trial. Contemp Clin Trials. 2023 Feb;125:107077. doi: 10.1016/j.cct.2022.107077. Epub 2022 Dec 30. PMID 36592818